CLINICAL TRIAL: NCT02079064
Title: Perioperative Effect of Desflurane Versus Total Intravenous Anesthesia With Propofol on Hemostasis Guided by Thromboelastometry in Splenectomy With Liver Cirrhosis.
Brief Title: Effects of Desflurane Versus Propofol on Hemostasis During Splenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Yasser Mostafa Samhan, Professor of Anesthesia, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Anesthesia 98T
Record Dates: First submitted 2014-02-27; First posted 2014-03-05 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2016-10

CONDITIONS: Status; Splenectomy
Keywords: Splenectomy; Desflurane; Propofol; TCI; ROTEM
MeSH Terms: interventions — Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desflurane (Experimental): Desflurane at 1 MAC and
  Interventions: Drug: Desflurane
- propofol (Experimental): propofol TCI (target controlled infusion) infusion of to keep a target plasma concentration between 2 and 5 µg ml-1
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Desflurane — Inhalational anesthetic
  Other Names: Suprane
  Arms: Desflurane
Drug: Propofol — Intravenous anesthetic that can be given by continuous infusion
  Other Names: Diprivan
  Arms: propofol

SUMMARY:
The aim of this prospective randomized study is to evaluate the perioperative effects of inhalational anesthesia (desflurane) and intravenous anesthesia (propofol) on hemostasis in patients undergoing splenectomy with liver cirrhosis guided by the new technology (ROTEM) and the traditional laboratory hemostatic markers.

DETAILED DESCRIPTION:
After obtaining approval from the Institutional Research Ethics Committee and informed written consent, thirty adult patients aged 25- 55 years of either sex, American Society of Anesthesiologists (ASA) class II- III (Child A) suffering from cytopenia scheduled for elective splenectomy will be recruited. Pancytopenia is defined as anemia (hemoglobin < 13.5 g/dL-male; <12 g/dL-female); leucopenia (total leukocyte count < 4,000/mm3) and thrombocytopenia (platelet count < 150,000/mm3). Child B and C, Hb < 10 g/dL platelet count < 50,000/mm3, White Blood Cells (WBCs) < 2,000/mm3, prothrombin time [PT] > 16 s and INR > 1.7, extremes of age, obese patients (body mass index >35 kg m-2), and those using oral anticoagulants, other antithrombotic drugs, or oral contraceptives, will be excluded from the study.

All patients will be premedicated with 0.05 mg kg-1 i.v midazolam half an hour before operation. In the operating room, continuous pulse oximetry, electrocardiogram, non-invasive arterial blood pressure, PECO2, end-tidal anesthetic agent, neuromuscular monitoring, core temperature (Infinity Kappa, Dräger, Lübeck, Germany) and hourly urine output will be monitored throughout the operation. Depth of anesthesia will be monitored by using Bispectral index (BIS). All IV fluids will be warmed, and a warm air blanket (Bair Hugger) will be applied to every patient.

Thirty eligible patients will be allocated randomly to one of two equal groups (15 patients each) according to a computer generated randomization list: group D; maintenance of anesthesia with inhaled desflurane at 1 minimum alveolar concentration (MAC); group P, maintenance of anesthesia with target-controlled infusion (TCI) propofol with a target plasma concentration of propofol between 2 and 5 µg ml-1. The concentration of volatile anesthetics or the rate of infusion of injected anesthetics will be titrated to maintain the BIS numerical value between 40-50.

Anesthesia will be induced in both groups using i.v. fentanyl 1.5- 2 µg kg-1 and propofol 2- 2.5 mg kg-1. Atracurium 0.5 mg kg-1 will be administered for neuromuscular block and continued according to the response to train-of-four peripheral nerve stimulation. After intubation, patients will be mechanically ventilated with 30% oxygen in air throughout surgery using a low flow system (1L min-1) to adjust an end-tidal carbon dioxide (PECO2) between 30- 35 mmHg. Acetated Ringer's solution will be given as a preload and maintenance at a rate of 5-7 ml kg-1 h-1. Patients' systolic arterial pressures will be maintained at 100 mmHg or 70% of the preoperative value, whichever is higher. Hypotension will be treated with i.v. crystalloid fluid loading or intravenous boluses of ephedrine as appropriate. No colloid transfusion will be allowed. Transfusions of red blood cells will be used to maintain hemoglobin levels equal to or above 8 g dl-1. Platelets or fresh frozen plasma will be infused only when indicated by ROTEM. At the end of surgery, neuromuscular blockade will be antagonized with 0.05 mg kg-1 neostigmine and 0.02 mg kg-1 atropine. Postoperative analgesia was provided by intravenous infusion of 1 gm acetaminophen and IV meperidine 1 mg kg-1 every 12 hours. Patients are given an anti-emetic ondansetron 4 mg postoperatively.

Blood Sampling:

Five blood samples will be collected; before operation, after ligation of splenic artery, immediate post-operative, 24 hours and three days after the operation. Each time, five ml of venous blood will be collected and assessment of the following parameters will be performed:

Complete blood picture:

1. Hemoglobin Concentration (by electronic cell counter).
2. Hematocrit (by electronic cell counter).
3. Platelet count (by electronic cell counter).
4. Red blood cells (by electronic cell counter).
5. White blood cells (by electronic cell counter).

Screening hemostatic tests:

1. Prothrombin Time (PT) (by conventional method).
2. International Normalized Ratio (INR) (by conventional method).
3. Partial Thromboplastin Time (PTT) (by conventional method).

Specific hemostatic tests:

1. Soluble platelet selectin (sP-selectin) [enzyme-linked immunosorbent assay (ELISA)].
2. Fibrinogen level (coagulation method).
3. D-dimer level (ELIZA).

At each sample time (0.3 ml blood) will be taken for measuring the following ROTEM variables:

* The time until initial fibrin formation (clotting time CT).
* The kinetics of fibrin formation and clot development (clot formation time (CFT) and α- angle).
* The ultimate strength and stability of the fibrin clot (maximum clot firmness MCF).
* Clot lysis (fibrinolysis). The previous parameters provide information about platelet activation, fibrin formation and clot retraction (all stages of the developing and resolving clot). Blood samples are activated extrinsically (by tissue factor) and intrinsically (by contact activator) via commercially available tests. Furthermore, fibrinogen levels will be assessed by measuring clot strength (MCF) in the presence of platelet inhibition (e.g., fib-TEM). This modified MCF represents the fibrin clot that developed in the absence of any platelets, i.e., the functional fibrinogen [6].

Routine laboratory tests:

1. Serum creatinine.
2. Alanine aminotransferase (ALT),aspartate aminotransferase (AST), albumin, bilirubin.

Routine investigations will be performed pre-, post-operative and on the third day.

Follow up of each patient will be done at out-patients clinic after one month to have thorough clinical examination, liver and kidney function tests, Child's Turcotte Pugh (CTP) score assessment, laboratory hematological tests and ROTEM assessment. This is important to assess post-operative complications, efficacy of splenectomy in improving cytopenia, and the influence of splenectomy on the natural course of disease.

Statistical Analysis:

No previous study was conducted to assess the effects of anesthetic agents on hemostasis during splenectomy with liver cirrhosis guided by ROTEM. Thus the calculation of the sample size is difficult and also the reagents required for ROTEM are expensive so we designed this thesis to be a pilot study. A sample size was chosen to be 15 patients in each group. Comparison between the two groups will be performed using Mann-Whitney test, while comparison within each group will be performed using Wilcoxon sign rank test. Comparison between repeated measures in both groups was performed using ANOVA. The data are considered significant if p values are ≤ 0.05. Statistical analysis will be performed with the aid of the Statistical Package for the Social Sciences (SPSS) computer program, version 12 windows (IBM, USA).

.

ELIGIBILITY:
Inclusion Criteria:

* Patient ASA physical status II and III.
* Age between 22-55 years.
* Child A suffering from pancytopenia.
* Type of surgery: splenectomy

Exclusion Criteria:

* Patients using oral anticoagulants
* Patients using antithrombotic drugs
* Patients using non steroidal anti-inflammatory drugs
* Patients using oral contraceptives
* Age less than 25 or more than 55 years
* Obese patients (body mass index >35 kg m-2)
* Pregnancy and lactation

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
maximum clot firmness (MCF) | Up to 1 month
  Ultimate strength and stability of the fibrin clot measured by ROTEM.

SECONDARY OUTCOMES:
clotting time CT | Up to 1 month
  The time until initial fibrin formation measured by ROTEM
clot formation time; CFT | Up to 1 month
  The kinetics of fibrin formation and clot development measured by ROTEM
D dimer | Up to 1 month
  Indication of coagulation and fibrinolysis
Platelet count | Up to 1 month
  Ability of clot formation
Prothrombin Time | Pre-operative, after ligation of splenic artery, immediate post-operative, 24 hours and three days after operation
  measures of the extrinsic pathway of coagulation
International Normalized Ratio (INR) | Pre-operative, after ligation of splenic artery, immediate post-operative, 24 hours and three days after operation
  measures of the extrinsic pathway of coagulation
sP-selectin | Pre-operative, after ligation of splenic artery, immediate post-operative, 24 hours and three days after operation
  Acts as a receptor that supports binding of leukocytes to activated platelets and endothelium.
Fibrinogen Level | Pre-operative, after ligation of splenic artery, immediate post-operative, 24 hours and three days after operation
  A soluble plasma glycoprotein, that is converted by thrombin into fibrin during blood clot formation
D-Dimer | Pre-operative, after ligation of splenic artery, immediate post-operative, 24 hours and three days after operation
  A fibrin degradation product (or FDP) present in the blood after a blood clot is degraded by fibrinolysis

CONTACTS AND LOCATIONS:
Overall Officials: Gehan G El-Fandy, M.D., Study Chair — Theodor Bilharz Research Institute
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Senzolo M, Burra P, Cholongitas E, Burroughs AK. New insights into the coagulopathy of liver disease and liver transplantation. World J Gastroenterol. 2006 Dec 28;12(48):7725-36. doi: 10.3748/wjg.v12.i48.7725. PMID 17203512
- [Result] Liangpunsakul S, Ulmer BJ, Chalasani N. Predictors and implications of severe hypersplenism in patients with cirrhosis. Am J Med Sci. 2003 Sep;326(3):111-6. doi: 10.1097/00000441-200309000-00001. PMID 14501224
- See also: Senzolo M, Burra P, Cholongitas E, Burroughs AK. New insights into the coagulopathy of liver disease and liver transplantation. World J Gastroenterol 2006; 12(48): 7725-36 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4087534/
- See also: Liangpunsakul S, Sithat M, Ulmer B, Chalasani. Predictors and implications of severe hypersplenism in patients with cirrhosis. Am J Med Sciences 2003; 326: 111-16. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Predictors+and+implications+of+severe+hypersplenism+in+patients+with+cirrhosis